CLINICAL TRIAL: NCT01769456
Title: Project PrEPare - An Open Label Demonstration Project and Phase II Safety Study of Pre-Exposure Prophylaxis Use Among 15 to 17 Year Old Young Men Who Have Sex With Men (YMSM) in the United States
Brief Title: An Open Label Demonstration Project and Phase II Safety Study of Pre-Exposure Prophylaxis Use Among 15 to 17 Year Old Young Men Who Have Sex With Men (YMSM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Gilead Sciences (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN 113 Version 2.0
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-11

CONDITIONS: HIV Infection
Keywords: HIV, PrEP, FTC/TDF, Truvada®
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PCC Behavioral Intervention Group (Experimental): PCC Behavioral Intervention combined with open label FTC/TDF (Truvada®) as PrEP
  Interventions: Behavioral: PCC; Drug: Emtricitabine/tenofovir (FTC/TDF (Truvada®))

INTERVENTIONS:
Behavioral: PCC — Personalized Cognitive Counseling (PCC) is based on the Model of Relapse Prevention and Gold's Self-Appraisal of Risk Behavior. PCC is a 1-hour, single-session, individual level intervention administered by a trained counselor in a clinic setting. Counselors ask the client to recall and describe a recent encounter of unprotected anal sex with another man of unknown or sero-discordant HIV status. The client then identifies and expresses thoughts, feelings, or attitudes that might have led to the high-risk behavior. The client and counselor examine and identify thoughts that may have led the client to decide to engage in high transmission risk sex. The client and counselor agree on strategies that can be used to deal with similar situations in the future.
  Other Names: Personalized Cognitive Counseling
Drug: Emtricitabine/tenofovir (FTC/TDF (Truvada®)) — All subjects will be provided with daily FTC/TDF (Truvada®) as Pre-exposure prophylaxis (PrEP) for 48 weeks.
  Other Names: FTC/TDF; Truvada®; Emtricitabine/tenofovir; PrEP

SUMMARY:
Approximately 100 HIV-uninfected YMSM at high risk of acquiring HIV infection, between the ages of 15 and 17 inclusive will be enrolled across all participating Adolescent Medicine Trial Units (AMTUs). Subjects will complete the behavioral intervention selected by all participating sites, Personalized Cognitive Counseling (PCC), and will then be provided with open label emtricitabine (FTC)/tenofovir (TDF) (Truvada®) as pre-exposure prophylaxis (PrEP). Behavioral and biomedical data will be collected at baseline and at 0, 4, 8, 12, 24, 36 and 48 weeks. Any subject who becomes HIV infected during the course of the study will be discontinued from the study agent and be followed for an additional 24 weeks after the study visit at which HIV infection is confirmed. Those subjects who meet specific bone or renal criteria at the Week 48 visit or the 24-Week HIV Seropositive visit will be followed for an additional 48 weeks in the Extension Phase to monitor longer-term outcomes of potential concerns.

DETAILED DESCRIPTION:
The aims of the study are to obtain additional data on the safety of FTC/TDF (Truvada®) and to evaluate acceptability, patterns of use, rates of adherence, and measured levels of drug exposure when YMSM are provided with open label FTC/TDF (Truvada®) and information regarding safety and efficacy of FTC/TDF (Truvada®) as PrEP based on prior studies in adults. The study will also examine patterns of sexual risk behavior among HIV-uninfected YMSM in the U.S. at high risk of acquiring HIV infection who are provided with open label FTC/TDF (Truvada®) as PrEP. The study will also explore the feasibility and acceptability of implementing an efficacious risk reduction behavioral intervention prior to the provision of PrEP- PCC. The inclusion of a behavioral intervention in this project not only addresses the ethical responsibility of providing at least the minimum risk reduction education to all subjects given the high HIV risk of the study population, but also builds behavioral skills to assist subjects in reducing their risk when not taking PrEP. Furthermore, the study will evaluate the process of protocol implementation to better understand how to best implement PrEP research and program practice at adolescent medicine sites, including an evaluation of consent procedures and the acceptability/feasibility of allowing youth minors to consent for their own participation in HIV prevention intervention, to the extent allowable by local laws and regulations, and to allow youth minor participation in a clinical trial without requiring disclosure of their sexual orientation and risk behaviors to their parents or legal guardians.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent;
* Male gender at birth;
* Age 15 years and 0 days through 17 years and 364 days, inclusive, at the time of signed informed consent;
* Self reports evidence of high risk for acquiring HIV infection including at least one of the following:

  * At least one episode of unprotected anal intercourse with an HIV-infected male partner or a male partner of unknown HIV status during the last 6 months;
  * Anal intercourse with 3 or more male sex partners during the last 6 months;
  * Exchange of money, gifts, shelter, or drugs for anal sex with a male partner during the last 6 months;
  * Sex with a male partner and has had a sexually transmitted infection (STI) during the last 6 months or at screening;
  * Sexual partner of an HIV-infected man with whom condoms were not consistently used in the last 6 months; or
  * At least one episode of anal intercourse where the condom broke or slipped off during the last 6 months;
* Tests HIV antibody negative at time of screening;
* Willing to provide locator information to study staff;
* Willing to take PrEP;
* Willing to participate in behavioral intervention;
* Reports intention not to relocate out of AMTU study area during the course of the study; and
* Does not have a job or other obligations that would require long absences from AMTU study area (greater than 4 weeks at a time).

Exclusion Criteria:

* Appears visibly distraught or presence of active serious psychiatric symptoms (e.g., active hallucinations, suicidal, homicidal, or exhibiting violent behavior) at the time of consent;
* Intoxicated or under the influence of alcohol or other drugs at the time of consent;
* Any significant uncontrolled, active or chronic disease process that, in the judgment of the site investigator, would make participation in the study inappropriate. (Appropriately managed conditions, like well-controlled diabetes, would not preclude enrollment; the site is encouraged to contact the Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 113 Protocol Team if they are having difficulty making the judgment.);
* History of bone fractures not explained by trauma;
* Acute or chronic hepatitis B infection as indicated by positive hepatitis B surface antigen (sAg) test at time of screening;
* Confirmed renal dysfunction (Creatinine Clearance (CrCl) < 75 ml/min calculated based on bedside Schwartz formula: Glomerular filtration rate (GFR) = (0.413 x (height in centimeters)) / (serum creatinine in mg/dl)), or serum creatinine > upper limit of normal (ULN), or history of renal parenchymal disease or presence of only one kidney at time of screening;
* Confirmed ≥ Grade 2 hypophosphatemia at time of screening;
* Confirmed ≥ Grade 2 hematologic system abnormality (White Blood Count (WBC), Absolute Neutrophil Count (ANC), hemoglobin, or platelets) at time of screening;
* Confirmed ≥ Grade 2 hepatobiliary system abnormality (Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), or bilirubin) at time of screening;
* Confirmed proteinuria as indicated by urine dipstick result ≥ 1+ at time of screening, regardless of urine protein to creatinine ratio (UP/C);
* UP/C > 0.37 g/g at time of screening, regardless of urine dipstick protein result;
* Confirmed normoglycemic glucosuria as indicated by urine dipstick result ≥ 1+ in the presence of normal serum glucose (<120 mg/dL) at time of screening;
* A confirmed Grade ≥ 3 toxicity on any screening evaluations;
* Known allergy/sensitivity to the study agent or its components;
* Concurrent participation in an HIV vaccine study or other investigational drug study, including oral or topical PrEP (microbicide) studies;
* Use of disallowed medications; or
* Inability to understand spoken English.

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, PhD, Study Chair — Stroger Hospital of Cook County
Locations (6):
- United States (6):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Colorado - The Children's Hospital of Denver, Aurora, Colorado
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - Fenway Institute, Boston, Massachusetts
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Hosek SG, Landovitz RJ, Kapogiannis B, Siberry GK, Rudy B, Rutledge B, Liu N, Harris DR, Mulligan K, Zimet G, Mayer KH, Anderson P, Kiser JJ, Lally M, Brothers J, Bojan K, Rooney J, Wilson CM. Safety and Feasibility of Antiretroviral Preexposure Prophylaxis for Adolescent Men Who Have Sex With Men Aged 15 to 17 Years in the United States. JAMA Pediatr. 2017 Nov 1;171(11):1063-1071. doi: 10.1001/jamapediatrics.2017.2007. PMID 28873128
- [Derived] Havens PL, Perumean-Chaney SE, Patki A, Cofield SS, Wilson CM, Liu N, Anderson PL, Landovitz RJ, Kapogiannis BG, Hosek SG, Mulligan K. Changes in Bone Mass After Discontinuation of Preexposure Prophylaxis With Tenofovir Disoproxil Fumarate/Emtricitabine in Young Men Who Have Sex With Men: Extension Phase Results of Adolescent Trials Network Protocols 110 and 113. Clin Infect Dis. 2020 Feb 3;70(4):687-691. doi: 10.1093/cid/ciz486. PMID 31179503
- See also: ATN website — http://www.atnonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This research was conducted at 6 clinical sites. Accrual was open between 7/16/2013 and 9/30/2014.
Groups:
- PCC Behavioral Intervention Group: PCC is based on the Model of Relapse Prevention and Gold's Self-Appraisal of Risk Behavior. The PCC intervention was conducted as a 1-hour, single-session, individual level intervention administered by a trained counselor in a clinic setting. After completion of the PCC intervention, all subjects were provided with daily FTC/TDF (Truvada®) as Pre-exposure prophylaxis (PrEP) for 48 weeks.
Period: Overall Study
Arm/Group | PCC Behavioral Intervention Group
Started | 78 (1 subject inadvertently enrolled, discontin'd after baseline, re-enrolled later and completed study)
Completed | 41
Not Completed | 37
Not completed — Lost to Follow-up | 19
Not completed — Withdrawal by Subject | 3
Not completed — Did not receive PCC intervention | 6
Not completed — Moved out of the area | 3
Not completed — No wk 0 visit w/in 30 days of screening | 5
Not completed — Parental request to youth to withdraw | 1

BASELINE CHARACTERISTICS:
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.52 (0.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Modified binary variable for race, distinguishing only those who identified as Black/African-American from those who did not.
  Participants
    Black/African-American: Black/African-American | 33
    Black/African-American: Non-Black/African-American | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Derived variable combining information on race and ethnicity.
  Participants
    Race/ethnicity: Asian/Pacific Islander | 2
    Race/ethnicity: Black/African American | 23
    Race/ethnicity: White | 11
    Race/ethnicity: White/Hispanic | 16
    Race/ethnicity: Other/Mixed Race | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78
Lumbar spine bone mineral density (BMD) [Mean (Standard Deviation); unit: g/cm2] — Population: Subjects with DXA data at baseline.
  g/cm2
    number analyzed (Participants) | 75
    (all) | 1.03 (0.15)
Femoral neck bone mineral density (BMD) [Mean (Standard Deviation); unit: g/cm2] — Population: Subjects with DXA data at baseline.
  g/cm2
    number analyzed (Participants) | 75
    (all) | 0.99 (0.16)
Total body bone mineral density (BMD) [Mean (Standard Deviation); unit: g/cm2] — Population: Subjects with DXA data at baseline.
  g/cm2
    number analyzed (Participants) | 75
    (all) | 1.15 (0.11)
Total hip bone mineral density (BMD) [Mean (Standard Deviation); unit: g/cm2] — Population: Subjects with DXA data at baseline.
  g/cm2
    number analyzed (Participants) | 75
    (all) | 1.06 (0.15)
Number of participants reporting unprotected sex with a male partner in the past month [Count of Participants; unit: Participants] — From the participant ACASI question referring to male partners in the past month:
  "Of these males, how many did you have unprotected oral or anal sex with in the past month?"
  An event is defined as an answer of greater than 0. Population: Participants who provided a response to this question on the ACASI survey.
  Participants
    number analyzed (Participants) | 60
    (all) | 52
Number of male sexual partners in the last month [Mean (Standard Deviation); unit: male sexual partners] — From the participant ACASI question:
  "During the past month, how many male partners have you had sexual contact with (oral or anal)?" Population: Participants who provided a response to this question on the ACASI survey.
  male sexual partners
    number analyzed (Participants) | 73
    (all) | 1.95 (2.15)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serum Creatinine Event of Grade 1 or Higher Over the Course of the Study
Description: This represents one of the indicators associated with the objective: Additional safety data regarding FTC/TDF (Truvada®) use among HIV-uninfected YMSM.
  Participants were assessed for any serum creatinine event of Grade 1 or higher over the course of the study (Week 0 through Week 48).
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- PCC Behavioral Intervention Group: PCC Behavioral Intervention Group combined with open label FTC/TDF (Truvada®) as PrEP
  PCC: Personalized Cognitive Counseling (PCC) is based on the Model of Relapse Prevention and Gold's Self-Appraisal of Risk Behavior. PCC is a 1-hour, single-session, individual level intervention administered by a trained counselor in a clinic setting.
  Emtricitabine/tenofovir (FTC/TDF (Truvada®)): All subjects will be provided with daily FTC/TDF (Truvada®) as Pre-exposure prophylaxis (PrEP
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 78
Participants | 0

2. Primary Outcome: Lumbar Spine Bone Mineral Density: Percent Change From Baseline to Week 48
Description: The percent change in lumbar spine BMD from baseline measurement to Week 48 is calculated as:
  Percent change= [(Value at Week 48 - Value at Baseline)/(Value at Baseline)] x 100
  This represents one of the indicators associated with the objective: Additional safety data regarding FTC/TDF (Truvada®) use among HIV-uninfected YMSM.
Time Frame: Baseline, Week 48
Population: Subjects with dual energy x-ray absorptiometry (DXA) data at both baseline and Week 48.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 43
percent change | 2.59 (3.22)
Statistical Analysis 1: Comparison: PCC Behavioral Intervention Group; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test — Reported p-value is the calculated value provided by SAS output

3. Primary Outcome: Femoral Neck Bone Mineral Density: Percent Change From Baseline to Week 48
Description: The percent change in femoral neck BMD from baseline measurement to Week 48 is calculated as:
  Percent change= [(Value at Week 48 - Value at Baseline)/(Value at Baseline)] x 100
  This represents one of the indicators associated with the objective: Additional safety data regarding FTC/TDF (Truvada®) use among HIV-uninfected YMSM.
Time Frame: Baseline, Week 48
Population: Subjects with DXA data at both baseline and Week 48.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 43
percent change | 1.16 (3.66)
Statistical Analysis 1: Comparison: PCC Behavioral Intervention Group; Test type: Other; p = 0.0236, Wilcoxon Signed Rank Test

4. Primary Outcome: Total Body Bone Mineral Density: Percent Change From Baseline to Week 48
Description: The percent change in total body BMD from baseline measurement to Week 48 is calculated as:
  Percent change= [(Value at Week 48 - Value at Baseline)/(Value at Baseline)] x 100
  This represents one of the indicators associated with the objective: Additional safety data regarding FTC/TDF (Truvada®) use among HIV-uninfected YMSM.
Time Frame: Baseline, Week 48
Population: Subjects with DXA data at both baseline and Week 48.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 43
percent change | 1.29 (2.28)
Statistical Analysis 1: Comparison: PCC Behavioral Intervention Group; Test type: Other; p = 0.0003, Wilcoxon Signed Rank Test

5. Primary Outcome: Total Hip Bone Mineral Density: Percent Change From Baseline to Week 48
Description: The percent change in total hip BMD from baseline measurement to Week 48 is calculated as:
  Percent change= [(Value at Week 48 - Value at Baseline)/(Value at Baseline)] x 100
  This represents one of the indicators associated with the objective: Additional safety data regarding FTC/TDF (Truvada®) use among HIV-uninfected YMSM.
Time Frame: Baseline, Week 48
Population: Subjects with DXA data at both baseline and Week 48.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 43
percent change | 1.27 (3.71)
Statistical Analysis 1: Comparison: PCC Behavioral Intervention Group; Test type: Other; p = 0.0236, Wilcoxon Signed Rank Test

6. Primary Outcome: Number of Participants With Decrease in Bone Mineral Density
Description: The proportion of subjects with DXA data through Week 48 who experienced varying degrees of decrease in absolute BMD in at least one region (spine, hip, or whole body).
  This represents one of the indicators associated with the objective: Additional safety data regarding FTC/TDF (Truvada®) use among HIV-uninfected YMSM.
Time Frame: 48 weeks
Population: Enrolled subjects with DXA results for baseline and Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 43
Participants
  Decrease in absolute BMD >=1% baseline to Wk48 | 16
  Decrease in absolute BMD >=5% baseline to Wk48 | 2
  Decrease in absolute BMD >10% baseline to Wk48 | 0

7. Primary Outcome: Behavioral Disinhibition/Risk Compensation: Number of Participants Reporting Unprotected Sex
Description: Behavioral disinhibition/risk compensation was assessed based on a number of questions, including the following related to unprotected sex from the participant ACASI:
  "Of these males [male partners], how many did you have unprotected oral or anal sex with since the last time you took this survey?" An event is defined as an answer of greater than 0.
  This represents one of the indicators associated with the objective: Additional safety data regarding FTC/TDF (Truvada®) use among HIV-uninfected YMSM.
Time Frame: Week 48
Population: Participants providing data for this question at Week 48.
Measure: Count of Participants; unit: Participants
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 31
Participants | 25

8. Primary Outcome: Behavioral Disinhibition/Risk Compensation: Number of Male Sexual Partners
Description: Behavioral disinhibition/risk compensation was assessed based on a number of questions, including the following related to related to number of male sexual partners from the participant ACASI:
  "Since the last time you took this survey, how many male partners have you had sexual contact with (oral or anal)?"
  This represents one of the indicators associated with the objective: Additional safety data regarding FTC/TDF (Truvada®) use among HIV-uninfected YMSM.
Time Frame: Week 48
Population: Participants providing data for this question at Week 48.
Measure: Mean (Standard Deviation); unit: male sexual partners
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 46
male sexual partners | 1.64 (1.88)

9. Primary Outcome: Acceptability of PrEP Regimen and Study Visits
Description: This represents one of the indicators associated with the objective: Acceptability when YMSM are provided open label FTC/TDF (Truvada®) and information regarding the safety and efficacy of PrEP from prior studies.
  Acceptability of PrEP as measured by the acceptability assessment that includes questions on usability of PrEP, user-friendliness of the medication regimen, including an assessment of side effects and delivery format, and acceptability of behavioral intervention sessions.
Time Frame: Week 12
Population: Enrolled subjects with Week 12 data (individual row totals vary based on number of subjects providing responses for each question)
Measure: Count of Participants; unit: Participants
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 62
Participants
  Size of the pill: number analyzed (Participants) | 59
  Size of the pill: Did not like it at all | 3
  Size of the pill: Did not like | 14
  Size of the pill: Liked | 36
  Size of the pill: Liked a lot | 6
  Taste of the pill: number analyzed (Participants) | 60
  Taste of the pill: Did not like it at all | 8
  Taste of the pill: Did not like | 27
  Taste of the pill: Liked | 22
  Taste of the pill: Liked a lot | 3
  Color of the pill: number analyzed (Participants) | 61
  Color of the pill: Did not like it at all | 2
  Color of the pill: Did not like | 8
  Color of the pill: Liked | 42
  Color of the pill: Liked a lot | 9
  Taking the pill every day: number analyzed (Participants) | 59
  Taking the pill every day: Did not like it at all | 1
  Taking the pill every day: Did not like | 17
  Taking the pill every day: Liked | 34
  Taking the pill every day: Liked a lot | 7
  Taking part in the study: Did not like it at all | 1
  Taking part in the study: Did not like | 0
  Taking part in the study: Liked | 26
  Taking part in the study: Liked a lot | 35
  HIV test at every visit: Did not like it at all | 1
  HIV test at every visit: Did not like | 4
  HIV test at every visit: Liked | 25
  HIV test at every visit: Liked a lot | 32
  Risk Reduction Counseling at every visit: number analyzed (Participants) | 61
  Risk Reduction Counseling at every visit: Did not like it at all | 2
  Risk Reduction Counseling at every visit: Did not like | 3
  Risk Reduction Counseling at every visit: Liked | 26
  Risk Reduction Counseling at every visit: Liked a lot | 30
  Questions about sexual behavior at every visit: Did not like it at all | 2
  Questions about sexual behavior at every visit: Did not like | 10
  Questions about sexual behavior at every visit: Liked | 36
  Questions about sexual behavior at every visit: Liked a lot | 14
  Physician exam by a doctor: number analyzed (Participants) | 60
  Physician exam by a doctor: Did not like it at all | 1
  Physician exam by a doctor: Did not like | 9
  Physician exam by a doctor: Liked | 35
  Physician exam by a doctor: Liked a lot | 15
  Health clinic for study visits: Did not like it at all | 1
  Health clinic for study visits: Did not like | 3
  Health clinic for study visits: Liked | 41
  Health clinic for study visits: Liked a lot | 17

10. Primary Outcome: Estimation of Medication Adherence by Dried Blood Spot (DBS) Results
Description: This outcome addresses the objective: Rates of adherence and measured levels of drug exposure when YMSM are provided open label FTC/TDF (Truvada®) and information regarding the safety and efficacy of PrEP from prior studies.
  Medication adherence is estimated by factors including levels of drug exposure as measured by DBS red blood cell (RBC) samples.
  The TFV dosing level was translated into number of dosing days per week for week 8 onwards using lab estimates as follows: '<2 days' is defined as <350 (fmol/punch), '2 days' as 350 to 700 (fmol/punch), '4 days' as >700 to 1250 (fmol/punch), and 'Daily' as >1250 (fmol/punch).
  The TFV dosing level was translated into number of dosing days for week 4 using lab estimates as follows: '<2 days' is defined as <275 (fmol/punch), '2 days' as 275 to 525 (fmol/punch), '4 days' as >525 to 950 (fmol/punch),and 'Daily' as >950 (fmol/punch)
Time Frame: Week 4, Week 12, Week 24, Week 36, Week 48
Population: Number analyzed in each row varies based on the number of enrolled subjects with DBS data available for each week.
Measure: Count of Participants; unit: Participants
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 78
Participants
  DBS RBC TFV-DP (fmol/punch), Week 4: number analyzed (Participants) | 65
  DBS RBC TFV-DP (fmol/punch), Week 4: Below level of quantification | 3
  DBS RBC TFV-DP (fmol/punch), Week 4: <2 days | 12
  DBS RBC TFV-DP (fmol/punch), Week 4: 2 days | 11
  DBS RBC TFV-DP (fmol/punch), Week 4: 4 days | 24
  DBS RBC TFV-DP (fmol/punch), Week 4: Daily | 15
  DBS RBC TFV-DP (fmol/punch), Week 8: number analyzed (Participants) | 63
  DBS RBC TFV-DP (fmol/punch), Week 8: Below level of quantification | 3
  DBS RBC TFV-DP (fmol/punch), Week 8: <2 days | 13
  DBS RBC TFV-DP (fmol/punch), Week 8: 2 days | 14
  DBS RBC TFV-DP (fmol/punch), Week 8: 4 days | 21
  DBS RBC TFV-DP (fmol/punch), Week 8: Daily | 12
  DBS RBC TFV-DP (fmol/punch), Week 12: number analyzed (Participants) | 60
  DBS RBC TFV-DP (fmol/punch), Week 12: Below level of quantification | 3
  DBS RBC TFV-DP (fmol/punch), Week 12: <2 days | 17
  DBS RBC TFV-DP (fmol/punch), Week 12: 2 days | 7
  DBS RBC TFV-DP (fmol/punch), Week 12: 4 days | 22
  DBS RBC TFV-DP (fmol/punch), Week 12: Daily | 11
  DBS RBC TFV-DP (fmol/punch), Week 24: number analyzed (Participants) | 55
  DBS RBC TFV-DP (fmol/punch), Week 24: Below level of quantification | 15
  DBS RBC TFV-DP (fmol/punch), Week 24: <2 days | 18
  DBS RBC TFV-DP (fmol/punch), Week 24: 2 days | 5
  DBS RBC TFV-DP (fmol/punch), Week 24: 4 days | 12
  DBS RBC TFV-DP (fmol/punch), Week 24: Daily | 5
  DBS RBC TFV-DP (fmol/punch), Week 36: number analyzed (Participants) | 44
  DBS RBC TFV-DP (fmol/punch), Week 36: Below level of quantification | 17
  DBS RBC TFV-DP (fmol/punch), Week 36: <2 days | 11
  DBS RBC TFV-DP (fmol/punch), Week 36: 2 days | 6
  DBS RBC TFV-DP (fmol/punch), Week 36: 4 days | 7
  DBS RBC TFV-DP (fmol/punch), Week 36: Daily | 3
  DBS RBC TFV-DP (fmol/punch), Week 48: number analyzed (Participants) | 40
  DBS RBC TFV-DP (fmol/punch), Week 48: Below level of quantification | 19
  DBS RBC TFV-DP (fmol/punch), Week 48: <2 days | 8
  DBS RBC TFV-DP (fmol/punch), Week 48: 2 days | 2
  DBS RBC TFV-DP (fmol/punch), Week 48: 4 days | 7
  DBS RBC TFV-DP (fmol/punch), Week 48: Daily | 4

11. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was session interesting, was it relevant to their life, and did they learn from the session)
Time Frame: 48 weeks
Population: Data not collected; only one type of risk reduction intervention was ultimately implemented.
Groups:
- PCC Behavioral Intervention Group: PCC Behavioral Intervention Group combined with open label FTC/TDF (Truvada®) as PrEP
  PCC: Personalized Cognitive Counseling (PCC) is based on the Model of Relapse Prevention and Gold's Self-Appraisal of Risk Behavior. PCC is a 1-hour, single-session, individual level intervention administered by a trained counselor in a clinic setting.
  Emtricitabine/tenofovir (FTC/TDF (Truvada®)): All subjects will be provided with daily FTC/TDF (Truvada®) as Pre-exposure prophylaxis (PrEP).
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants Using Text Messaging Reminders
Description: This represents one of the indicators associated with the objective: Acceptability and feasibility of text message reminders.
Time Frame: Baseline through Week 48
Population: The analysis population for those discontinued is the population (N=22) of those who initially signed up to receive reminders.
Measure: Count of Participants; unit: Participants
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 78
Participants
  Signed up for text message reminders | 22
  Discontinued reminders while on study agent: number analyzed (Participants) | 22
  Discontinued reminders while on study agent | 2
  Discontinued reminders while still on study: number analyzed (Participants) | 22
  Discontinued reminders while still on study | 1

13. Secondary Outcome: Rating of the Reasons for Missing Medications on a 4-point Likert Scale.
Description: This represents one of the indicators associated with the objective: Acceptability and feasibility of text message reminders, as measured by subject rating of the reasons for missing medications on a 4-point Likert scale.
  Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
Time Frame: 48 weeks
Population: Enrolled subjects with a Week 48 visit; individual rows may have varying Ns due to the number of subjects providing data for each question.
Measure: Count of Participants; unit: Participants
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 46
Participants
  Were away from home: number analyzed (Participants) | 40
  Were away from home: Never | 15
  Were away from home: Rarely | 8
  Were away from home: Sometimes | 12
  Were away from home: Often | 5
  Were too busy with other things: number analyzed (Participants) | 40
  Were too busy with other things: Never | 15
  Were too busy with other things: Rarely | 10
  Were too busy with other things: Sometimes | 7
  Were too busy with other things: Often | 8
  Simply forgot: number analyzed (Participants) | 40
  Simply forgot: Never | 21
  Simply forgot: Rarely | 4
  Simply forgot: Sometimes | 7
  Simply forgot: Often | 8
  Had too many study pills to take: number analyzed (Participants) | 40
  Had too many study pills to take: Never | 36
  Had too many study pills to take: Rarely | 4
  Had too many study pills to take: Sometimes | 0
  Had too many study pills to take: Often | 0
  Wanted to avoid side effects: number analyzed (Participants) | 40
  Wanted to avoid side effects: Never | 37
  Wanted to avoid side effects: Rarely | 2
  Wanted to avoid side effects: Sometimes | 1
  Wanted to avoid side effects: Often | 0
  Did not want others to notice you taking meds: number analyzed (Participants) | 40
  Did not want others to notice you taking meds: Never | 36
  Did not want others to notice you taking meds: Rarely | 3
  Did not want others to notice you taking meds: Sometimes | 0
  Did not want others to notice you taking meds: Often | 1
  Had a change in daily routine: number analyzed (Participants) | 40
  Had a change in daily routine: Never | 27
  Had a change in daily routine: Rarely | 4
  Had a change in daily routine: Sometimes | 5
  Had a change in daily routine: Often | 4

14. Secondary Outcome: Demographic and/or Behavioral Difference Between Study Groups. Behavioral Disinhibition/Risk Compensation Endpoints Will be Compared.
Time Frame: 48 weeks
Population: Data were not collected.
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 0

15. Secondary Outcome: Evaluation of the Process of Protocol Implementation
Description: Brief phone interviews and review of written institutional review board (IRB) correspondence will be conducted for all sites whether the study is approved at that site or not. If approved, the steps needed for approval and how barriers were addressed will be examined. If the study was rejected, the reasons for disapproval, the IRB's interpretation of the risk of PrEP, and other barriers will be examined. In addition, data from a survey specific to each site's IRB's responses of minor YMSM inclusion in PrEP studies will be evaluated.
  NOTE: Data collected to address this outcome were primarily qualitative in nature, and as such are not presented here. For more information on this outcome, refer to:
  Gilbert AL, Knopf AS, Fortenberry JD, Hosek SG, Kapogiannis BG, Zimet GD. Adolescent Self-Consent for Biomedical Human Immunodeficiency Virus Prevention Research. J Adolesc Health. 2015 Jul;57(1):113-9.
Time Frame: 48 weeks
Population: Quantitative data were not collected for this outcome.
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 0

16. Secondary Outcome: Demographic and/or Behavioral Differences Between Youth Who Are Interested in Participating in a PrEP Study Versus Those Who Are Not.
Description: Behavioral disinhibition/risk compensation endpoints will be compared.
Time Frame: 48 weeks
Population: Data were not collected.
Arm/Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of the study, from the start of enrollment on 7/16/2013 until the completion of subject follow-up on 8/18/2016 (approximately 3 years).
Description: Per protocol, only grade 3 and higher clinical adverse events and lab toxicities are systematically recorded on the Adverse Event Evaluation Form and reported here.
Arm/Group | PCC Behavioral Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 3/78
Other Adverse Events (participants affected / at risk) | 6/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCC Behavioral Intervention Group (N=78)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCC Behavioral Intervention Group (N=78)
Weight Decreased (Investigations) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions Publication Policy outlines procedures for the development and review of abstracts, publications, and presentations. The Adolescent Medicine Leadership Group (AMLG) retains custody of and primary rights to the data. Use of data must be approved by the protocol team and AMLG.